CLINICAL TRIAL: NCT05737485
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study, in Healthy Adult Participants and Open-Label Single Ascending Dose Study in Adults With Primary Ciliary Dyskinesia Caused by Pathogenic Mutations in the DNAI1 Gene to Evaluate the Safety and Tolerability of RCT1100
Brief Title: Study Evaluating the Safety and Tolerability of RCT1100 in Healthy and PCD Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReCode Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCT1100-101
Record Dates: First submitted 2023-01-20; First posted 2023-02-21 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Primary Ciliary Dyskinesia; PCD; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RCT1100 (Experimental): Drug: RCT1100 single dose
  Interventions: Drug: RCT1100

INTERVENTIONS:
Drug: RCT1100 — RCT1100 mRNA therapy supplied as varying dose strengths administered via oral inhalation using nebulizer

SUMMARY:
This is the first-in-human study with RCT1100 and is designed to provide initial safety and tolerability data for future clinical studies.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and tolerability of a single ascending dose of inhaled RCT1100 administered via nebulizer to healthy participants and patients with Primary Ciliary Dyskinesia caused by a pathogenic mutation in the DNAI1 Gene.

ELIGIBILITY:
Major Inclusion Criteria:

* Healthy, adult, male or female of, 18-75 years of age, inclusive, at screening.
* Participant has disease causing mutations in the DNAI1 gene
* The participant has a forced expiratory volume in one second (FEV1) of at least 50% predicted.

Major Exclusion Criteria:

* History or presence of clinically significant medical, surgical, clinical laboratory, or psychiatric condition or disease.
* History of cancer, with exception of adequately treated basal cell or squamous cell carcinoma of the skin.
* Medically significant hemoptysis
* Anticoagulation therapy for the treatment of a pulmonary embolus or has had a pulmonary embolus in the last 6 months of screening.
* Active tuberculosis infection.
* Laboratory abnormalities in clinical laboratory tests at screening:

  1. Serum creatinine level
  2. Total bilirubin, aspartate aminotransferase or alanine aminotransferase values
  3. Hematological or coagulation values outside the normal reference range
* Any medical history of disease that has the potential to cause a rise in total bilirubin over the ULN
* History of alcohol abuse or drug addiction with the last year of screening.
* Active smoker (vaping included).

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
The number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs). | From Baseline Through Day 180
  Safety and tolerability as assessed by number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs), as well as an adverse event of special interest (AESI): "Fever", which will include body temperature and any associated symptoms (chills, myalgia).

CONTACTS AND LOCATIONS:
Overall Officials: John Matthews, MBBS, MCRP, PhD, Study Chair — ReCode Therapeutics, Inc.
Locations (4):
- PPD - Las Vegas Research Unit, Las Vegas, Nevada, United States
- Macquarie University, Sydney, New South Wales, Australia
- New Zealand Clinical Research, Auckland, New Zealand
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No